CLINICAL TRIAL: NCT07278310
Title: STAR Trial (Siegel Transcatheter Aortic Valve Replacement in Patients With Symptomatic Severe Aortic Stenosis)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MiRus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MR-002
Record Dates: First submitted 2025-12-02; First posted 2025-12-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Symptomatic Severe Native Aortic Stenosis; Aortic Stenosis
Keywords: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Investigational Device- Siegel TAVR
  Interventions: Device: Siegel TAVR Device
- Control Arm (Active Comparator): Commercially available TAVR device- Sapien TAVR or Evolute TAVR
  Interventions: Device: TAVR Device

INTERVENTIONS:
Device: TAVR Device — Commercially available TAVR Device
  Arms: Control Arm
Device: Siegel TAVR Device — Siegel TAVR Device
  Arms: Treatment Arm

SUMMARY:
To evaluate the safety and efficacy of Siegel™ TAVR System in the treatment of subjects with symptomatic severe native aortic stenosis.

DETAILED DESCRIPTION:
The primary objective is to assess the acute and long-term safety and efficacy of the Siegel THV device in adult subjects with symptomatic, severe native calcific aortic stenosis eligible for the transcatheter aortic valve replacement.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for entry in this study if ALL the following conditions are met:

1. Age ≥ 18 years
2. Symptomatic, severe native calcific aortic stenosis in subjects at low, intermediate or high surgical risk AVA ≤ 1.0 cm2 or AVA index ≤ 0.6 cm2/m2 or Jet velocity ≥ 4.0 m/s or mean gradient ≥ 40 mmHg or dimensionless Index <0.25
3. New York Heart Association Functional Class ≥ 2
4. Requires aortic valve replacement and is indicated for TAVR as determined by the Heart Team (composed of an experienced interventional cardiologist and an experienced cardiac surgeon)
5. Eligible for transfemoral delivery of a TAVR
6. Native aortic annulus suitable for safe placement of Siegel 23mm, transcatheter heart valve. Preprocedural measurements by TTE and CT of aortic annulus area (330- 440 mm2 )
7. Understands the study requirements and the treatment procedures and provides written informed consent
8. Subject agrees to complete all required scheduled follow-up visits.

Exclusion Criteria:

Subjects will be excluded for entry in this study if ANY of the following conditions are met:

Anatomical

1. Cardiac anatomy precluding safe placement of a transcatheter aortic valve.
2. Iliofemoral anatomy (vessel diameter < 5.5mm) precluding safe placement of commercially available transcatheter aortic valves (SAPIEN 3 or Evolut).
3. Pre-existing prosthetic heart valve or ring except in the mitral position.
4. Unicuspid aortic valve
5. Severe aortic regurgitation (>3+)
6. Severe mitral or severe tricuspid regurgitation(>3+) requiring intervention.
7. Moderate to severe mitral stenosis.
8. Hypertrophic obstructive cardiomyopathy (HOCM)
9. Echocardiographic evidence of intracardiac mass, thrombus or vegetation requiring treatment.
10. Significant aortic disease including abdominal aortic or thoracic aneurysm defined as maximal luminal diameter 5.5 cm or greater or ascending aortic aneurysm defined as maximal luminal diameter 5 cm or greater.

    Clinical
11. Evidence of an acute myocardial infarction ≤ 30 days before enrollment.
12. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to the index procedure
13. Blood dyscrasias as defined: leukopenia (WBC < 3000 cell/mL, anemia (Hgb < 9 g/dL), thrombocytopenia (platelet count < 50,000 cells/mL), history of bleeding diathesis or coagulopathy.
14. Untreated clinically significant Coronary Artery Disease (CAD) requiring revascularization
15. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support within the past 30 days.
16. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical heart assistance within 30 days of enrollment
17. Need for emergency surgery for any reason
18. Ventricular dysfunction with left ventricular ejection fraction (LVEF) < 25% as measured by resting echocardiogram
19. Recent (within 6 months) cerebrovascular accident (CVA) or transient ischemic attack (TIA).
20. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 30 days of enrollment
21. Renal insufficiency (eGFR < 30 ml/min per the Cockcroft-Gault formula) and/or renal replacement therapy, or end stage renal disease requiring chronic dialysis
22. GI bleeding within the past 3 months
23. Severe lung disease (FEV1 < 50% predicted) or currently on home oxygen
24. History of cirrhosis or any active liver disease
25. Significant abdominal or thoracic aortic disease (such as porcelain aorta, abdominal aortic aneurysm > 5.0 cm, severe calcification, aortic coarctation, etc.) that would preclude safe passage of the delivery system
26. Severe pulmonary hypertension (e.g., PA systolic pressure ≥ 2/3 systemic pressure)
27. A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated: aspirin, heparin, ticlopidine and clopidogrel, contrast media, nickel, cobalt ,chromium, titanium, molybdenum, rhenium, polyethylene materials.
28. Ongoing sepsis, including active endocarditis
29. BMI > 50 kg/m2
30. Subject refuses a blood transfusion
31. Life expectancy < 12 months due to associated non-cardiac co-morbid conditions
32. Other medical, social, or psychological conditions that in the opinion of an Investigator precludes the subject from appropriate consent
33. Severe dementia (resulting in either inability to provide informed consent for the trial/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits)
34. Currently participating in an investigational drug or another investigational device trial
35. Subject is contraindicated for cardiac CT
36. Subject belongs to a vulnerable population (Vulnerable subject populations are defined as individuals with mental disability, persons in nursing homes, children, impoverished persons, homeless persons, nomads, refugees, and those permanently incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1025 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality, all stroke and cardiovascular rehospitalization | 1 Year
  The primary endpoint is the composite of all-cause mortality, all stroke, and cardiovascular rehospitalization (valve-related or procedure-related per VARC-3) at 1 year.

IPD SHARING:
Plan to Share IPD: No